CLINICAL TRIAL: NCT07400081
Title: Effectiveness of a Community-based Intervention Programme to Promote Well-being in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group Polyclinics (Other Government)
Collaborators: Lien Foundation (Unknown); Institute of Mental Health, Singapore (Other); Lee Kong Chian School of Medicine, Nanyang Technological University (Unknown); Fei Yue Community Services (Unknown); Club HEAL (Unknown)
Responsible Party: Principal Investigator, Chua Yu Cong, Eugene, Family Physician, Consultant, National Healthcare Group Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-1289
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Well-being/Quality of Life; Mental Health
Keywords: Community-based intervention; Well-being; Older adults; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Community-based intervention through structured psychoeducation and social prescription
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Waitlist Control
- Intervention (Other): Community-based Intervention
  Interventions: Behavioral: Community-based Intervention

INTERVENTIONS:
Behavioral: Community-based Intervention — Psychoeducation Programme
  Arms: Intervention

SUMMARY:
This study is conducted to assess the effectiveness of a community intervention programme on improving well-being, levels of distress, and loneliness in older adults (aged 55 years old and above), who have symptoms of depression.

Social Service Agencies (SSAs) will conduct focal talks on well-being for the community. As part of the focal talks, the Public Health Questionnaire-9 (PHQ-9) will be conducted. Attendees with a PHQ-9 score of 1-9 will be invited to take part in the study. Up to 300 participants will be recruited and randomised into 2 arms: control arm (150 participants) and intervention arm (150 participants).

Participants in the intervention arm will undergo 8-week community intervention programme which includes 4 sessions on well-being and continuous follow-up with a Health Companion. Participants in the control arm will be offered to join a programme conducted by the SSAs 8 weeks after recruitment into the study. The programmes offered to the control group are independent of the study.

DETAILED DESCRIPTION:
Study Procedures:

Control arm: Participants randomised into the control arm will not be offered any programmes for 8 weeks after their recruitment into the study. After 8 weeks, the SSAs will offer the participants an intervention programme that is independent of the study.

Intervention arm: Participant in the intervention arm will undergo 4 face-to-face, group psychoeducation sessions, conducted fortnightly over a period of 8 weeks. The sessions will teach the participants about well-being and share with them strategies to improve their well-being. Health Companions from the SSAs will conduct check-ins with the participants over the phone, and recommend some nearby activities for them.

Methods and assessments:

Questionnaires including the 6-item De Jong Gierveld Loneliness Scale, Warwick-Edinburgh Mental Wellbeing Scale, Patient Health Questionnaire-9, and Generalised Anxiety Disorder-7 at the baseline and endpoint for all participants.

Expected risks:

During the administration of the questionnaires, participants may feel uncomfortable or upset. Participants may choose to refuse to asnwer any of the questions, or take a break at any time during the questionnaire administration.

Participants in the intervention arm may feel discomfort, anxiousness or distress while undergoing the intervention programme. Participants may cease their enrolment in the study, or be encouraged to attend clinical follow-ups or reach out to the Social Service Agencies' Community Intervention Team (COMIT).

Safety Review Plan:

As this study does not involve any invasive procedures, the study team does not foresee any adverse events related to the study.

Data Quality Assurance:

The PI or study team member will review all data collection forms on an ongoing basis for data completeness, accuracy and protocol compliance, after every data collection timepoint.

Data entry and storage:

For hardcopy data, they will be stored in designated locked cabinet(s) or room(s) that are accessible to authorized study personnel only. For electronic data, they will be stored on in a secured computer that is password protected. The databases will not contain subject identifiers and the data linking subject identifiers and the subject identification codes will be stored separately.

Sample size calculation:

An a priori power analysis was conducted to determine the required sample size for detecting a statistically significant difference in the primary outcome, the Warwick-Edinburgh Mental Well-being Scale (WEMWBS), between the intervention and control arms. The effect size based on standardised mean differences (SMD) for this calculation was informed by a comprehensive systematic review by Blodgett et al. (2022), which reported a medium to large range of SMD from 0.38 to 0.72 for selected themes and subthemes of intervention across studies. To ensure the study is adequately powered for a conservative estimate, the smallest effect size from this range, d = 0.38, was used for the calculation. The power analysis was performed for a two-tailed independent samples t-test using the pwr package in R, with a standard significance level (α) of 0.05 and a desired power (1-β) of 0.80. The results indicated that a minimum of 110 participants per group is required. To account for a potential 20% attrition rate, the minimum recruitment target is about 130 participants per arm. The study team rounded up the number to 150 participants per arm, with a total of 300 participants to be recruited.

Statistical and analytical plans:

Data will be analysed using SPSS/Stata/R. Normality of the data will be checked using the Kolmogorov-Smirnov test. Differences between variables will be tested by t-test and Mann-Whitney U test for normal and non-normal continuous variables, respectively and chi-square test or Fisher-exact test for categorical variables. Associations with the improvement in scores will be analysed via multivariable regressions. P value <0.05 will indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 and above
* Score of 1-9 on the PHQ-9 questionnaire
* Able to speak and understand English, Chinese or Malay
* Able to provide informed consent
* Be willing to use common technologies (such as phone calls, texting via SMS/whatsapp) for communication

Exclusion Criteria:

* PHQ-9 score of 0
* PHQ-9 score of 10 or more
* Actively being followed up by a mental health professional
* On psychotropic medication or are undergoing psychotherapy
* Have other mental disorders or are suicidal
* Have physical difficulties, cognitive impairment or difficulties with speech, sight and hearing or mobility that may prevent their engagement in activities

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Well-being | 8 weeks
  Measured by Warwick-Edinburgh Mental Well-being Scale (WEMWBS)

SECONDARY OUTCOMES:
Depressive symptoms | 8 weeks
  Measured by Patient Health Questionnaire-9 (PHQ-9)
Anxiety symptoms | 8 weeks
  Measured by Generalised Anxiety Disorder-7 (GAD-7)
Loneliness | 8 weeks
  Measured by De Jong Gierveld Loneliness Scale

OTHER OUTCOMES:
Acceptability, feasibility and satisfaction of the intervention | 8 weeks
  Measured through qualitative interviews

CONTACTS AND LOCATIONS:
Locations (1):
- National Healthcare Group Polyclinics, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No